CLINICAL TRIAL: NCT00997932
Title: A Pilot Study of Early Postpartum Intrauterine Contraception
Acronym: ImmPPIUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Gretchen Stuart, MD, MD, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SFP3-14
Record Dates: First submitted 2009-09-28; First posted 2009-10-20 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Unplanned Pregnancy
Keywords: levonorgestrel releasing intrauterine device; levonorgestrel releasing intrauterine contraception; unintended pregnancy prevention; postpartum contraception
MeSH Terms: interventions — Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Complete Cohort (Other): The complete cohort of all women enrolled and stated they wanted an LNG-IUS between 48 and 72 hours of vaginal delivery.
  Interventions: Drug: Levonorgestrel-Releasing Intrauterine Contraceptive System (LNG-IUS), 52 Mg, 5 Year Duration

INTERVENTIONS:
Drug: Levonorgestrel-Releasing Intrauterine Contraceptive System (LNG-IUS), 52 Mg, 5 Year Duration — Levonorgestrel-Releasing Intrauterine Contraceptive System, 52 Mg, 5 Year Duration Postpartum placement of LNG-IUS within 10 minutes - 48 hours
  Other Names: LNG-IUS

SUMMARY:
This is a prospective clinical trial of ultrasound guided intrauterine contraception insertion 10 minutes - 48 hours after vaginal delivery of single infant. A six month follow-up will entail three follow-up visits; 4-6 weeks, 3 months, and 6 months.

The objective of this study is to measure intrauterine device (IUD) expulsion and the feasibility of conducting a future clinical trial to evaluate placement of the levonorgestrel-releasing intrauterine contraceptive 10 minutes - 48 hours postpartum.

DETAILED DESCRIPTION:
This was a single arm cohort study of women who desired to receive a levonorgestrel releasing intrauterine system (LNG-IUS) within 48 hours of uncomplicated vaginal delivery.

Women were enrolled during a prenatal care visit when they reported they desired to use the LNG-IUS after the birth of their infant.

Forty women stated enrolled in the study prior to labor, and baseline data were obtained. After delivery 29 women remained both interested in the study and were still eligible to receive the LNG-IUS prior to discharge from the hospital.

Of the 29 women who received the LNG-IUS prior to discharge from the hospital 11 women had an LNG-IUS expulsion prior to 6 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant with a single gestation of at least 27 completed weeks estimated gestational age, with no complications of pregnancy including, but not limited to, preeclampsia, non-gestational diabetes, anemia.
* Desires to use intrauterine contraception (IUD) after delivery
* Anticipates having a vaginal delivery
* No intention to leave the area 7 months after enrollment
* Able to consent to participate in the study in English
* Has no known uterine anomalies
* Has no allergies to any components of the intrauterine contraception

Exclusion Criteria:

* Prior cesarean delivery
* Having been treated for pelvic inflammatory disease within 3 months prior to the start of the pregnancy
* Allergic to betadine
* Allergy to lidocaine
* Medical or personal conditions which in the judgment of study staff contradict participation in the study
* Any contraindications to use of the levonorgestrel-releasing intrauterine contraceptive system which includes: known or suspected breast carcinoma, acute liver disease or liver tumor, history of ectopic pregnancy, cervical cancer or carcinoma in situ
* After enrollment, and after delivery of the infant but before IUD insertion subjects will be excluded by checking with the attending obstetric physician and/or obstetric medical chart for the following:

  * Endometritis or chorioamnionitis during the intrapartum period
  * Membranes ruptured for greater than 24 hours prior to delivery
  * Fever greater than or equal to 38C
  * The need to use additional medications other than pitocin and/or misoprostol to control postpartum bleeding

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Stuart, MD, MPHTM, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All women enrolled who stated they wanted an IUD postpartum. Of those 40 enrolled, 29 were eligible, and did receive, the IUD prior to discharge from the hospital.
Groups:
- Immediate Insertion: Women in the immediate insertion arm received a Mirena intrauterine contraceptive system within 10 minutes and up to 48 hours of delivery.
  Mirena Intrauterine Contraceptive System: Postpartum placement of the IUD within 10 minutes - 48 hours
Period: Overall Study
Arm/Group | Immediate Insertion
Started | 29
Completed | 27
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Immediate Insertion
Number analyzed (Participants) | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The results are presented for the 29 women who received the IUD. Baseline data are presented for the 29 women who received the IUD and the 11 women who did not.
  years | 23 [21 to 29]
Sex: Female, Male [Count of Participants; unit: Participants] — females only because this was a female contraception study Population: All women enrolled who stated they wanted an IUD postpartum. Of those 40 enrolled, 29 were eligible, and did receive, the IUD prior to discharge from the hospital.
  Participants
    Female | 29
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race White Black Other Hispanic ethnicity Population: All women enrolled who stated they wanted an IUD postpartum. Of those 40 enrolled, 29 were eligible, and did receive, the IUD prior to discharge from the hospital.
  Participants
    Race: White | 17
    Race: Black | 9
    Race: Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
Previous contraceptive use, marital status, employment, [Count of Participants; unit: Participants] — Population: All women enrolled who stated they wanted an IUD postpartum. Of those 40 enrolled, 29 were eligible, and did receive, the IUD prior to discharge from the hospital.
  Participants
    Employed: Yes | 2
    Employed: No | 27
    Married or Cohabitating: Yes | 9
    Married or Cohabitating: No | 20
    Prior use of contraception: Yes | 29
    Prior use of contraception: No | 0

OUTCOME MEASURES:

1. Primary Outcome: IUD Expulsion
Description: Expulsion of the LNG-IUS
Time Frame: From time of insertion to final study date which is 6 months after IUD insertion.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Insertion
Number analyzed (Participants) | 29
Participants | 11

ADVERSE EVENTS:
Groups:
- No IUD Insertion: Women in this group underwent baseline data collection, stated they would like to enroll and receive an IUD between 10 minutes and 48 hours postpartum. These women were not eligible to receive the IUD due to delivery elsewhere, medical complications in peri-partum period.
Arm/Group | Immediate Insertion | No IUD Insertion
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/11
Other Adverse Events (participants affected / at risk) | 0/29 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No